CLINICAL TRIAL: NCT00397579
Title: Therapy Targeting the Interleukin-3 Receptor (IL3R) for Patients With Relapsed or Refractory and Elderly or Poor-Risk Acute Myeloid Leukemia (AML) or High-Risk Myelodysplastic Syndrome With DTIL3 (IND# 11314): a Phase I/II Clinical Trial
Brief Title: DT388IL3 Fusion Protein in Treating Patients With Acute Myeloid Leukemia or Myelodysplastic Syndromes
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU 012013-061
Record Dates: First submitted 2006-11-08; First posted 2006-11-09 (Estimated); Results first posted 2019-04-23 (Actual); Last update posted 2019-04-23 (Actual); Status verified 2019-03

CONDITIONS: Leukemia; Myelodysplastic Syndromes; Blastic Plasmacytoid Dendritic Cell Neoplasm
Keywords: adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(15;17)(q22;q12); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); recurrent adult acute myeloid leukemia; secondary acute myeloid leukemia; untreated adult acute myeloid leukemia; de novo myelodysplastic syndromes; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes; blastic plasmacytoid dendritic cell neoplasm; plasmacytoid dendritic cell leukemia; CD123+
MeSH Terms: conditions — Leukemia; Myelodysplastic Syndromes; Blastic Plasmacytoid Dendritic Cell Neoplasm; Congenital Abnormalities; Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- SL-401 (Experimental): Patients will be treated with a maximum of five doses of approximately 15min IV infusions of DT388IL3/SL-401 over a ten day period at a maximum of once daily.
  Interventions: Drug: DT388IL3

INTERVENTIONS:
Drug: DT388IL3 — Intravenously via a 3 cc plastic syringe as a 15 minute bolus infusion daily for five days.

SUMMARY:
RATIONALE: Combinations of biological substances in DT388IL3 fusion protein may be able to carry cancer killing substances directly to the cancer cells.

PURPOSE: This phase I/II trial is studying the side effects and best dose of DT388IL3 fusion protein and to see how well it works in treating patients with acute myeloid leukemia or myelodysplastic syndromes.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of DT_388IL3 fusion protein in patients with refractory or relapsed or poor-risk acute myeloid leukemia (AML) or high-risk myelodysplastic syndromes (MDS).
* Define the dose-limiting toxicities of this regimen in these patients.
* Measure the pharmacokinetics of this regimen in these patients.
* Measure the immune responses in patients treated with this regimen.
* Evaluate response and correlate with disease type (relapsed/refractory or poor-risk de novo AML or high-risk MDS), pretreatment marrow blast percentage, and leukemia blast interleukin-3 receptor density.

OUTLINE: This is a phase I, multicenter, dose-escalation study followed by a phase II, open-label study.

* Phase I: Patients receive DT_388IL3 IV over 15 minutes daily for 5 days in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of DT_388IL3 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

* Phase II: An additional 15 patients receive DT_388IL3 at the MTD as in phase I. Patients undergo serum and blast collection periodically for laboratory studies, including analysis of expression of interleukin-3 receptors and anti-DT_388IL3 antibodies at baseline. Samples are also analyzed by immunoenzyme assays and flow cytometry.

After completion of study treatment, patients are followed periodically for up to 5 years.

PROJECTED ACCRUAL: A total of 50 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of 1 of the following:

  * Histologically or morphologically confirmed acute myeloid leukemia (AML), meeting 1 of the following criteria:

    * Relapsed or refractory AML after treatment with ≥ 1 prior conventional induction therapy

      * Patients in early first relapse must not have a matched donor available and/or be ineligible for allogeneic stem cell transplantation
    * Poor-risk AML, as defined by any of the following criteria:

      * Treatment-related AML, unless associated with favorable cytogenetics (e.g., inversion 16, t[16;16], t[8;21], t[15;17]), and ineligible for stem cell transplantation
      * Antecedent hematological disease (e.g., myelodysplastic syndromes, myelofibrosis, or polycythemia vera) that evolved to AML (≥ 20% blasts) and ineligible for stem cell transplantation
      * De novo AML (must be > 70 years of age)
      * AML with unfavorable cytogenetics (e.g., abnormalities of chromosomes -7, -5, 7q-, or 5q-; complex [≥ 3] abnormalities; or abnormalities of 11q23, excluding t[9;11], t[9;22], inversion 3, t[3;3], and t[6;9]), regardless of age, and ineligible for allogeneic stem cell transplantation
  * High-risk myelodysplastic syndromes diagnosed by morphologic, histochemical, or cell surface marker criteria

    * Resistant or intolerant to chemotherapy
    * Ineligible for or unwilling to undergo immediate allogeneic stem cell transplantation
* Bone marrow index (i.e., percent cellularity × percent blasts) ≤ 40% at time of treatment
* No active CNS leukemia

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Bilirubin ≤ 1.5 mg/dL
* ALT and AST < 2.5 times upper limit of normal
* Albumin ≥ 3 mg/dL
* Creatinine ≤ 1.5 mg/dL
* LVEF ≥ 50%
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 2 weeks after completion of study treatment
* No complicated medical or psychiatric problems that would preclude study compliance
* No concurrent serious uncontrolled infection or disseminated intravascular coagulation
* No myocardial infarction within the past 6 months
* No allergies to diphtheria toxin
* No requirement for oxygen

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No other concurrent antineoplastic drugs
* No concurrent radiotherapy
* No concurrent corticosteroids as antiemetics
* No concurrent hematopoietic growth factors (e.g., epoetin alfa, interleukin-11, filgrastim [G-CSF], or sargramostim [GM-CSF])
* No concurrent intravenous immunoglobins

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2013-05; Primary Completion 2017-07-27 (Actual); Study Completion 2017-07-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arthur E. Frankel, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

REFERENCES:
- [Derived] Frankel AE, Woo JH, Ahn C, Pemmaraju N, Medeiros BC, Carraway HE, Frankfurt O, Forman SJ, Yang XA, Konopleva M, Garnache-Ottou F, Angelot-Delettre F, Brooks C, Szarek M, Rowinsky E. Activity of SL-401, a targeted therapy directed to interleukin-3 receptor, in blastic plasmacytoid dendritic cell neoplasm patients. Blood. 2014 Jul 17;124(3):385-92. doi: 10.1182/blood-2014-04-566737. Epub 2014 May 23. PMID 24859366

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | SL-401
Started | 11
Completed | 11
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Patients with BPDCN treated with SL-401.
Arm/Group | SL-401
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 10
Age, Continuous [Mean (Full Range); unit: years] | 68 [40 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 11
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (CR+PR+SD): Percentage of Participants Experiencing Response
Description: Patients will be treated with a maximum of five doses of approximately 15min IV infusions of DT388IL3/SL-401 over a ten day period at a maximum of once daily.
  Response to Treatment will be evaluated as follows:
  Complete response (CR): patient has a normal whole blood count; platelets with absent blasts in peripheral blood or marrow; no evidence of nodal involvement or liver/spleen involvement; no skin lesion involvement.
  Partial Response (PR); patient experiences a decrease of 50% or more in marrow blasts and skin lesions; and there is a decrease in the size of the nodes/liver/spleen.
  Stable Disease (SD); failure to achieve at least PR, and there is no evidence of progression for 2 months.
  Failure: death during treatment or disease progression characterized by an increase in the percentage bone marrow blast or an increase in skin or node/liver or spleen size.
  Reported is the percentage of participants experiencing either CR, PR or SD.
Time Frame: From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 2 months
Measure: Number; unit: percentage of participants
Arm/Group | SL-401
Number analyzed (Participants) | 11
percentage of participants | 81.8

ADVERSE EVENTS:
Time Frame: 10 days
Arm/Group | SL-401
All-Cause Mortality (participants affected / at risk) | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 11/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SL-401 (N=11)
AST (Hepatobiliary disorders) | 4 (4)
Neutropenia (Blood and lymphatic system disorders) | 1 (1)
ALT (Hepatobiliary disorders) | 3 (3)
Thrombocytopenia (Blood and lymphatic system disorders) | 4 (4)
Hyponatremia (Blood and lymphatic system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-11-22): https://cdn.clinicaltrials.gov/large-docs/79/NCT00397579/Prot_SAP_000.pdf